CLINICAL TRIAL: NCT01573260
Title: Tango for Treatment of Motor and Non-motor Manifestations in Parkinson's Disease: A Randomized Control Study.
Brief Title: Tango for Treatment of Motor and Non-motor Manifestations in Parkinson's Disease.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Ron Postuma, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEN-11-261
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Tango
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Argentinean Tango (Experimental): A biweekly class of argentinean tango for a period of 3-months the intervention for this arm
  Interventions: Other: Argentinean Tango classes
- A 'wait-list' control group (Placebo Comparator): Intervention: Patient will receive information about exercise in PD. After 12 weeks, these patients will then start the same 12-weeks tango program.
  Interventions: Other: Simple pamphlet about the exercise in PD

INTERVENTIONS:
Other: Argentinean Tango classes — Tango participants will attend an 1-hour Argentinean Tango classes twice a week during 12 weeks, with experienced professional tango instructors.
  Arms: Argentinean Tango
Other: Simple pamphlet about the exercise in PD — Controls will follow their usual schedule of pharmacological treatment; will be provided by simple pamphlet about the exercise in PD, and will otherwise to go about their lives as usual.
  Arms: A 'wait-list' control group

SUMMARY:
Parkinson's disease involves many motor difficulties as well as non-motor ones. Recent research has strongly suggested that exercise is very important for Parkinson's disease. We are interested especially in dance as a form of exercise, because it combines physical movements with balance tasks, social engagement, and mental stimulation. Therefore, we think dance classes may be a very beneficial exercise for Parkinson's disease; the purpose of this study is to see if Argentinean Tango classes might improve motor and non-motor manifestations of Parkinson's disease.

DETAILED DESCRIPTION:
There is accumulating evidence for positive effects of exercise on gait speed, strength, balance, and quality of life for people with PD. Habitual physical activity can lower risk for developing PD. In toxin-induced animal models of PD, exercise may decrease neuronal injury. The key components of an exercise program in PD include: 1) cueing strategies to improve gait; 2) cognitive movement strategies to improve transfers; 3) exercises to improve balance, and 4) training of joint mobility and muscle power to physical capacity. Traditional exercise programs can meet these needs but often they are not very appealing for older adults including patients with PD. Unfortunately more than half of individuals with PD does not meet the recommended daily level physical activity.

There is a connection between music and level of Dopamine, which is pivotal for establishing and maintaining behavior. According to recent study music-induced emotional states can increase dopamine release, partially explaining how musical experiences are so valued and why music is an especially potent pleasurable stimulus for most people, and is frequently used to affect emotional states.

The development of interventions which combine exercise, with accessibility, enjoyability, good motivation to practice regularly improving mood and stimulating cognition would be ideal for individuals with PD. Dance may provide all of these characteristics, and so may be an affective useful and accessible intervention to improve motor impairments. Dance requires dynamic balance and permanent adjustment to the environment at the same time. It promotes enjoyment and encouragement interest in continuing participation. Habitual social dancers have superior balance, gait function, and reaction times compared with age-matched nondancers. Regular dancing improves balance and functional mobility, and increases motivation to continue healthful exercise-related behaviours in older adults.

There is also evidence that exercise has a positive impact on cognitive function in vulnerable populations. Musical exercise improved cognitive function in residents of long- term care facilitations without diagnosis of dementia and in patients with established Alzheimer's disease. Particularly dance produces clinically important changes in measures of mental status and behaviour in patients with moderate to severe dementia.

Social isolation is an important cause of the development of depression in the older population and it may be caused by numbers of factors, including mobility limitations: medical illness, and economic difficulties. The relationship between social isolation and depression is clear, as is the link between social engagement and improved mood and perceived quality of life. There is also an important link between social disengagement, depression and cognitive decline in elderly population. Dance classes occur in a group setting and it is forced social interaction, which may produce noticeable improvement in mood and subsequently decrease cognitive decline.

There is currently an insufficient body of literature on dance for PD and much additional work is needed. Most studies on dance in PD have used small sample sizes and assessed short-term effects and long-term effects of dance intervention only focused in motor manifestations of PD. Consequently, the effect of dance on cognition, mood and motivation has not been yet explored in PD. There is insufficient literature about what type of dance is more beneficial for motor and non-motor manifestations in PD.

Why Argentinean tango?

Better improvements of balance and complex gait were observed in elderly participants in tango lessons compared with a walking group. Beneficial effect of Argentine tango was also suggested, compared to traditional exercise for improving balance and functional mobility in patients with PD. Furthermore, a positron emission tomography (PET) study has shown increased activity in the basal ganglia when tango movements were performed with a metered and predictable beat. Tango requires particular motor skills, including frequent initiation and cessation, a variety of movement speeds, rhythmic variation, and spontaneous multidirectional perturbations. These features target motor impairments with movement initiation, turning, and bradykinesia. Interesting, tango could also effectively address freezing of gait (FOG), because some step patterns mimic the rehabilitation exercises designed for those with FOG. Visual cues, such as a foot to step over, can improve FOG. Tango technique which involve stepping over a partner's foot, tapping a partner's foot, or crossing one foot over another, are steps similar to conventional rehabilitation for FOG. In addition, tango involves rhythmic rocking, or alternating shift of center of mass from foot to foot, which can be another good strategy for freezing. Tango appeared to have a larger effect on freezing compared to other styles of dancing (waltz/foxtrot). Tango involves the practicing of control of movement speed and size, which may improve walking velocity and stride length. It also adds slow and quick steps of varying lengths and requires continual adjustment of these features. Tango may be especially beneficial for addressing backward walking, a critical area given the tendency for falls in the backward direction in PD6. Surprisingly in a recent study, tango even significantly improved upper extremity function, which it may be reflective of a global impact of exercise on bradykinesia. Better improvements of balance and complex gait were observed in elderly participants in tango lessons compared with a walking group. No studies have examined the effect of tango on cognitive function, mood and motivation in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for inclusion if they have a diagnosis of idiopathic PD.
* The subjects must speak either English or French sufficiently to fill out questionnaires and understand the instructions for dance classes (classes will be bilingual).

Exclusion Criteria:

1. Patients who cannot stand for at least 30 min and walk for ≥3 m without an assistive device.
2. Individuals with Hoehn and Yahr stage IV- V (severe and nonambulatory)
3. Dementia, defined according to PD dementia criteria as MMSE< 26/30 and ADL impairment secondary to cognitive loss, or inability to understand consent process60
4. Serious hearing and vision problems that could affect the participation in dance classes.
5. Change to dopaminergic therapy over the preceding three months, or changes to antiparkinsonian medication are anticipated during the study protocol
6. Serious medical conditions, including cardiac disease or evidence of musculoskeletal problem which precludes dancing or can be worsened by exercise
7. History of frequent falls, with more than 3 falls in the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Postuma, MD, Principal Investigator — Montreal General Hospital
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886

RESULTS

PARTICIPANT FLOW:
Groups:
- Argentinean Tango: A biweekly 3-month tango program
  Argentinean Tango classes: Tango participants will attend an 1-hour Argentinean Tango classes twice a week during 12 weeks, with experienced professional tango instructors.
- A 'Wait-list' Control Group: Patient information about exercise in PD. After 12 weeks, these patients will then start the same 12-weeks tango program.
  Simple pamphlet about the exercise in PD: Controls will follow their usual schedule of pharmacological treatment; will be provided by simple pamphlet about the exercise in PD, and will otherwise to go about their lives as usual.
Period: Overall Study
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Started | 18 | 15
Completed | 18 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Tango | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (8.1) | 63.2 (9.9) | 63.7 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 7 | 12 | 19
Disease duration [Mean (Standard Deviation); unit: years] | 7.7 (4.6) | 5.5 (4.4) | 6.5 (4.49)

OUTCOME MEASURES:

1. Primary Outcome: Severity of PD (Unified Parkinson Disease Rating Scale - UPDRS, 2008 Version)
Description: This is the standard scale used for grading severity of PD. It starts with a patient self-administered questionnaire covering activities of daily living, motor symptoms, and non-motor domains. It also includes a systematic rated clinical interview assessing cognitive and psychiatric symptoms and motor complications of disease. A Hoehn and Yahr scale (5-point overall disease severity index) is included. Finally, there is a formal examination component (Part III) (performed in the medication 'on' state for this study). Total score for Unified Parkinson Disease Rating Scale is the sum of six subscales, ranging from 0 (best possible outcome) to 60 (worst possible symptoms)
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Number analyzed (Participants) | 18 | 15
units on a scale
  baseline | 24.7 (9.6) | 30.5 (13.6)
  follow-up | 24.4 (10.8) | 30.2 (12.0)

2. Secondary Outcome: MiniBESTest
Description: Balance will be assessed using a 14-item tool measuring performance of dynamic balance tasks. This test has high interrater and test-retest reliability in PD (intraclass correlation coefficient ≥ .92 and intraclass correlation coefficient ≥.88 respectively). Total score for MiniBESTest is the sum of foursubscales, ranging from 0 (worst possible balance) to 28 (best possible balance). Lower scores indicate greater deficits in balance. Two items have right and left assessment in which the lower score is used within the total score (directions specify which to use). For research, we used of both left and right data, thus calculating data based on 32 (vs 28) points.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Number analyzed (Participants) | 18 | 15
units on a scale
  Baseline | 28.3 (2.3) | 27.1 (3.9)
  Follow-up | 28.8 (0.4) | 26.0 (4.3)

3. Secondary Outcome: Number of Participants With a Fall in the Past 3 Months Using the Falls Questionnaire From the Canadian Longitudinal Study of Aging
Description: Falls will be assessed using an adapted version of the falls questionnaire from the Canadian Longitudinal Study of Aging focusing on the past 3 months. This questionnaire includes 2 questions to assess if the participants felt during the past year and then it assess if this fall happened within the last 3 months. If a participant answered 'yes' to both questions, then the participant screened positive for this outcome. In the results section, we reported the number of participant who answered 'Yes' to both questions.
Time Frame: 26 weeks
Measure: Number; unit: participants
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Number analyzed (Participants) | 18 | 15
participants | 0 | 1

4. Secondary Outcome: Freezing of Gait Questionnare (FOG_Q)
Description: Freezing of gait will be assessed using the Freezing of Gait Questionnare (FOG_Q), a 6-item tool measuring walking and freezing episodes. Higher scores indicate greater difficulty with walking and freezing. Six items each scored from 0 to 6 were summed to obtain the total score, ranging from 0 (best possible outcome) to 36 (worst possible outcome).
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Number analyzed (Participants) | 18 | 15
units on a scale
  Baseline | 2.0 (2.5) | 4.6 (5.9)
  Follow-up | 2.7 (3.8) | 4.1 (4.2)

5. Secondary Outcome: The Purdue Pegboard
Description: The Purdue Pegboard, a test of dexterity and speed in the hands will be assessed over 1 minute. We calculate the number of pins correctly placed on the board in a minute.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: correct pins per 60 sec
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Number analyzed (Participants) | 18 | 15
correct pins per 60 sec
  Baseline | 14.4 (2.0) | 13.1 (2.9)
  Follow-up | 13.8 (2.4) | 12.5 (3.1)

6. Secondary Outcome: The Montreal Cognitive Assessment
Description: This tool was designed to screen for mild cognitive impairment. This includes visuospatial tests (clock drawing, trail making, cube copying), confrontation naming, attention (digit span, backwards digit span, "A" test, sentence repetition), tests of verbal fluency, abstraction, short term memory, and orientation. Recently, it has been used widely in PD, and demonstrates excellent sensitivity for subtle cognitive deficits. Alternate versions (7.1 to 7.3, with a randomly-distributed order) will be administered to prevent training effects. Total score for the MoCA is the sum of eight subscales, ranging from 0 (worst possible outcome) to 30 (best possible symptoms)"
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Number analyzed (Participants) | 18 | 15
score
  Baseline | 27.0 (2.4) | 26.7 (2.8)
  Follow-up | 27.4 (2.1) | 26.1 (3.2)

7. Secondary Outcome: The Beck Depression Inventory (BDI)
Description: The BDI is a self-administered scale of 21 items (scored 0-3) which assesses depression symptoms. The Beck Inventory is one of the most commonly-used scales for depression in PD, and a recent consensus panel of the Movement Disorders Society concluded it was a scale of first choice for assessing depression in PD. Total score for the BDI is the sum of 21 items, ranging from 0 (best possible outcome) to 63 (worst possible symptoms)"
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Number analyzed (Participants) | 18 | 15
score
  Baseline | 7.9 (6.6) | 7.7 (5.3)
  Follow-up | 7.7 (7.2) | 7.3 (4.4)

8. Secondary Outcome: Apathy Evaluation Scale (AES)
Description: This is a 14-item patient-rated scale which measures cognitive, emotional, and behavioural symptoms of apathy. All items are rated on a 0 to 3 Likert Scale. The original 18-item scale has been shortened by four items, and wording simplified and it was reported to have excellent psychometric properties in PD (internal consistency reliability = 0.76, test-retest 1 week r = 0.90). Total score is ranging from 0 (best possible outcome) to 42 (worst possible symptoms).
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Number analyzed (Participants) | 18 | 15
score
  Baseline | 28.9 (7.3) | 26.8 (7.6)
  Follow-up | 31.3 (4.5) | 29.4 (5.9)

9. Secondary Outcome: The Krupp Fatigue Severity Scale
Description: The fatigue severity scale measures impact of fatigue with a 9-item questionnaire, with a 7-point Likert scale for each question It has been validated, and has been used in PD studies. Total score is ranging from 0 (best possible outcome) to 63 (worst possible fatigue).
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Number analyzed (Participants) | 18 | 15
score
  Baseline | 34.3 (12.2) | 33.3 (14.2)
  Follow-up | 30.8 (15.3) | 35.9 (11.9)

10. Secondary Outcome: The Parkinson's Disease Questionnaire is a Quality of Life(PDQ-39)
Description: The PDQ-39 is a quality of life index for PD. It consists of a 39-item questionnaire that asks about the impact of PD on a person's motor function, gait, mood, cognition, and activities of daily living. Patients are asked to indicate the frequency of each event by selecting one of 5 options: never/occasionally/sometimes/often/always or cannot do at all. Total score is ranging from 0 (best possible outcome) to 156 (worst possible quality of life).
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Number analyzed (Participants) | 18 | 15
score
  Baseline | 26.8 (17.1) | 25.8 (15.1)
  Follow-up | 26.4 (18.9) | 24.5 (12.9)

11. Secondary Outcome: Adherence to Treatment
Description: Compliance with dance therapy will be conducted by reconfirming the regular assistance to the dance sessions at week 12, to compare how many sessions were attended by the participants. The dance instructors will keep the track of dance classes' assistance.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Number analyzed (Participants) | 18 | 15
participants | 6 | 0

12. Secondary Outcome: Clinical Global Impression of Change
Description: Completed by both the examiner and the patient, the scale is a single question" Since you have enrolled in the study, how has your Parkinson's disease changed?". It will be scored as very much improved (6), much improved (5), minimally improved (4), no change (3), minimally worse (2), much worse (1), or very much worse(0).
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Number analyzed (Participants) | 18 | 15
units on a scale | 3.4 (1.3) | 3 (1)

13. Secondary Outcome: Exit Questionnaire
Description: An exit questionnaire ranking level of enjoyment and overall satisfaction with their dance/exercise program, scored from 1 (strongly agree) to 5 (strongly disagree), with open questions about willingness continuing practicing tango.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Number analyzed (Participants) | 18 | 15
units on a scale
  Finding tango or exercise enjoyable | 1.1 (0.3) | 2.1 (0.9)
  Feeling overall satisfaction | 1.1 (0.3) | 2 (0.8)

14. Secondary Outcome: Adverse Events
Description: Adverse events will be queried week 12 through a semi structured interview querying increase in falls, fatigue, pain, cramps or pain, in addition to open-ended questions regarding other potential adverse events. Events will be rated by the patient and investigator as mild, moderate, or serious. All serious adverse events will be reported to the research ethics board
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Number analyzed (Participants) | 18 | 15
percentage of participants | 22 | 13

ADVERSE EVENTS:
Arm/Group | Argentinean Tango | A 'Wait-list' Control Group
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15
Other Adverse Events (participants affected / at risk) | 4/18 | 2/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Argentinean Tango (N=18) | A 'Wait-list' Control Group (N=15)
Falls (Musculoskeletal and connective tissue disorders) | 2 | 2 — Falls
respiratory infection (Infections and infestations) | 1 | 0
mild fatigue and muscle cramps (Musculoskeletal and connective tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This was a relatively small study, and many of our negative results could be related to inadequate power. The higher baseline activity rate in the controls may have affected responsiveness to change.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No